CLINICAL TRIAL: NCT02518009
Title: Phenotype Modulations Following Treatment With Contrary Sex Hormones
Brief Title: GEnder Dysphoria Treatment in Sweden
Acronym: GETS
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Thomas Gustafsson Assoc Prof, PhD, MD, Karolinska Institutet
Other Study IDs: KI GETS
Record Dates: First submitted 2015-05-12; First posted 2015-08-07 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Transsexualism
MeSH Terms: conditions — Transsexualism | interventions — Estrogens; Androgens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples from blood, skin, muscle and fat
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Men with gender dysphoria: Genetic men treated with estrogen
  Interventions: Other: Genetic men treated with estrogen
- Women with gender dysphoria: Genetic women treated with androgen
  Interventions: Other: Genetic women treated with androgen

INTERVENTIONS:
Other: Genetic men treated with estrogen — Observational during estrogen treatment
  Groups: Men with gender dysphoria
Other: Genetic women treated with androgen — Observational during androgen treatment
  Groups: Women with gender dysphoria

SUMMARY:
Gender dysphoria (DSM-5) or transsexualism (ICD10) is a condition in which a person's feeling of gender identity is not congruent with the physical body. The hormonal treatment includes inhibition of one's own sex hormone production followed by treatment with testosterone or estrogen levels that are normal for the opposite sex. Seen as experimental model, this is a process that provides an opportunity to study the sex hormone dependent influences that explain differences in morbidity in men and women respectively. The differences that are especially significant but not well known is 1) metabolic changes in the regulation of glucose homeostasis and lipid metabolism 2) regulation of vascular function and structural effects on the heart and arteries 3) regulation of skeletal muscle mass and fat tissue 4) morphological and functional effects on discrete areas of the brain.

Therefore, the investigators will follow these patients for a year to study how the heart, blood vessels, brain, and risk factors for cardiovascular disease affected by altered sex hormone patterns and studying what happens in the muscles and fat in both the short and long term with respect to particular gene expression and epigenetic changes and link it to metabolic changes and body composition.

DETAILED DESCRIPTION:
At the Centre for andrology and sexual medicine at Karolinska University Hospital about 30 genetic males (MtF) and 25 genetic females (FtM) every year start hormone replacement therapy. This hormonal treatment includes inhibition of one's own sex hormone production (down regulation of the gonadal axis) followed by treatment with testosterone or estrogen levels that are normal for the opposite sex. Seen as experimental model, this is a process that provides an opportunity to study the sex hormone dependent influences that explain differences in morbidity in men and women respectively. Furthermore, the constitutional differences distinguish them from those that are dynamically addressable through change in the hormonal milieu. The differences that are especially significant but not well known is 1) metabolic changes in the regulation of glucose homeostasis and lipid metabolism 2) regulation of vascular function and structural effects on the heart and arteries 3) regulation of skeletal muscle mass and fat tissue 4) morphological and functional effects on discrete areas of the brain.

It is well known that testosterone has a dose-response effect on body composition in men while conditions are less well known in women. Thus, it is not known how the adult woman's body responds to male levels of testosterone, and if the dose response relation is similar or different than that of men. The clinical impression is that women have less effect of androgen on muscle mass than men. Furthermore, it is not known whether the qualitative properties are comparable, i.e. muscle force/unit area. The basic hypothesis is that there are no constitutional sex differences in androgen response. If there are differences, we are looking to identify differences in gene expression. Another hypothetical regulatory mechanism is epigenetic differences which are not dynamically modifiable by androgen exposition. Difference in cardiovascular morbidity between men and women is well known, but there is considerable confusion if and how radical changes of sex hormone levels affects the function of the cardiovascular system both with acute and chronic exposure. Radical change of estrogen and testosterone levels can also affect the risk for metabolic disorders (lipid, carbohydrate and protein metabolism) which can cause hazard for both metabolic diseases such as diabetes and cardiovascular disease in the long term but also be a risk for future muscle weakness and osteoporosis. Effects on the central nervous system as a result of changes of sex hormone profile are not well known. However, we have several observations indicating that changes in sex hormone levels have visual effects (shown by MRI and PET) on distinctive features of the central nervous system.

Therefore, we will follow these patients for a year to study how the heart, blood vessels, brain, and risk factors for cardiovascular disease affected by altered sex hormone patterns and studying what happens in the muscles and fat in both the short and long term with respect to particular gene expression and epigenetic changes and link it to metabolic changes and body composition. Forty volunteers with gender dysphoria, 20 MtF and 20 FtM, are studied before the onset of sex hormone therapy, after a four-week shutdown of endogenous sex hormones and during one year of sex hormone treatment.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy

Exclusion Criteria:

* Infectious disease
* Treatment with Warfarin or other anti coagulants.
* History of cardiovascular disease.
* Serious illness or mental disorder.
* Diabetes type 1
* Language difficulties

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects that are under investigation for gender dysphoria that have been accepted but not yet started their treatment with contrary sex hormones are asked if they want to participate.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Physiological changes in peripheral tissues | 5 years
  Expression level and changes in epigenetics in skeletal muscle, skin and adipose tissue and associate to metabolism, insulin sensitivity, muscle strength, adipokines and adipose tissue morphology changes and body composition.

SECONDARY OUTCOMES:
Arterial stiffness, endothelial function and structural and functional effects of the heart | 5 years
Regulation of skeletal muscle mass and fat tissue with effect on body composition | 5 years
Systemic immune system changes | 5 years
Metabolic changes in the regulation of glucose homeostasis and lipid metabolism | 5 years
Morphological and functional effects on discrete areas of the brain | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Wiik, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Subramanian N, Wiik A, Rullman E, Melin M, Lundberg TR, Flanagan J, Holmberg M, Dekanski A, Dhejne C, Arver S, Gustafsson T, Laurencikiene J, Andersson DP. Adipokine secretion and lipolysis following gender-affirming treatment in transgender individuals. J Endocrinol Invest. 2024 Sep;47(9):2249-2260. doi: 10.1007/s40618-024-02323-4. Epub 2024 Mar 9. PMID 38460092
- [Derived] Wiik A, Lundberg TR, Rullman E, Andersson DP, Holmberg M, Mandic M, Brismar TB, Dahlqvist Leinhard O, Chanpen S, Flanagan JN, Arver S, Gustafsson T. Muscle Strength, Size, and Composition Following 12 Months of Gender-affirming Treatment in Transgender Individuals. J Clin Endocrinol Metab. 2020 Mar 1;105(3):dgz247. doi: 10.1210/clinem/dgz247. PMID 31794605